CLINICAL TRIAL: NCT01650506
Title: Phase I Study of Erlotinib and Metformin in Triple Negative Breast Cancer
Brief Title: Study of Erlotinib and Metformin in Triple Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Kevin Kalinsky, Assistant Professor of Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAF3743
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: Triple Negative; Basal-like
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Erlotinib + Metformin (Experimental): This is a single arm phase 1 study. All patients will receive erlotinib and metformin.
  Interventions: Drug: Metformin; Drug: Erlotinib

INTERVENTIONS:
Drug: Metformin — Due to frequent GI upset in patients starting metformin the dose will be titrated up to the assigned dose level. The first metformin dose level will be 850 mg twice daily and be escalated to its maximum FDA approved dose of 850 mg three times daily. Dose escalation will follow the standard 3 + 3 design. Dose limiting toxicities will be determined during the first 5 weeks of therapy.
  Other Names: Glucophage
Drug: Erlotinib — Erlotinib dosing will start and remain at 150 mg daily.
  Other Names: Tarceva

SUMMARY:
Extended phase 1 trial of combined metformin and erlotinib in advanced triple negative breast cancer patients. The goals of the study are to establish the maximum tolerated combined dosing of erlotinib and metformin as well as deciding if there is a potential clinical utility of the combination in treating patients with triple negative breast cancer.

DETAILED DESCRIPTION:
Breast cancer has several different subtypes based upon measurement of expression of proteins found on the surface of the cancer cells. Cancers that lack expression of three of these proteins, namely the estrogen receptor, progesterone receptor, and human epidermal growth factor receptor 2 (HER2), are termed triple negative. By studying the molecular attributes of breast cancer cells from a large group of breast cancer patients, a profile of markers enriched in triple negative breast cancers (TNBC) was discovered. This profile includes loss of expression of the protein, Phosphatase and Tensin homolog (PTEN), increased expression of the protein, epidermal growth factor receptor (EGFR), and disruption of the cells ability to repair DNA. These alterations also allow the tumor to thrive and likely evade treatment. Observation has been made that the drug combination of metformin and erlotinib can inhibit triple negative cells with these alterations. A clinical trial will be conducted to test the ability of patients to tolerate the treatment (Phase I trial). This trial will be available to triple negative breast cancer patients with metastatic disease. Other goals of the study will be to confirm that the drugs are working properly and whether or not there are enough responses to the treatment to warrant additional studies. If the treatment proves to be effective, even if only in a subset of triple negative patients, future studies will focus on validating biomarkers that can identify patients that will respond to the drug combination, as well as discovering how cells become resistant to the treatment. The research has the potential to advance a new effective treatment for a highly lethal disease and thus could prolong patient survivals while maintaining a high quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pathologic diagnosis of triple negative breast cancer, OR Prior diagnosis of ER or P-R positive breast cancer [HER2 negative] that is demonstrated to be both ER and P-R negative (no or rare staining) on the patient's most recent biopsy.
* Patients with measurable or non-measurable metastatic disease (RECIST 1.1).
* At least one prior treatment for metastatic disease.
* Availability of adequate tumor tissue for exploratory analysis and plan to obtain the material.
* Patients must have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. No chemotherapy or radiotherapy may be given within 2 weeks prior to the start of protocol treatment.
* Patients must be ≥ 18 and < 80 years old.
* Performance Status: Eastern Cooperative Oncology Group (ECOG) 0-2.
* Life expectancy of greater than 12 weeks.
* Patients must have recovered from uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia.
* Required Laboratory Values: Absolute neutrophil count (ANC) ≥1,250/mm3, platelets ≥75,000/mm3, hemoglobin ≥8.5 g/dL, total bilirubin ≤1.5 x ULN, Aspartate Aminotransferase (AST)/Alanine Aminotransferase (ALT) ≤3.0 x ULN, alkaline phosphatase ≤2.5 x ULN, Patients must have either a normal serum creatinine (<= IULN) OR estimated creatinine clearance ≥ 60 ml/min (Cockcroft-Gault formula) within 14 days prior to registration.
* Concomitant Medications: Erlotinib is primarily metabolized by CYP3A4. Patients CANNOT be receiving enzyme-inducing or enzyme inhibiting agents listed here: Inhibitors: Amiodarone, Amprenavir, Atazanavir, Chloramphenicol, Clarithromycin, Conivaptan, Cyclosporine, Darunavir, Dasatinib, Delavirdine, Diltiazem, Erythromycin, Fluconazole, Fluoxetine, Fluvoxamine, Fosamprenavir, Imatinib, Indinavir, Isoniazid, Itraconazole, Ketoconazole, Lapatinib, Miconazole, Nefazodone, Nelfinavir, Posaconazole, Ritonavir, Quinupristin, Saquinavir, Tamoxifen, Telithromycin, Troleandomycin, Verapamil, Voriconazole. Inducers: Aminoglutethimide, Bexarotene, Bosentan, Carbamazepine, Efavirenz, Fosphenytoin, Griseofulvin, Modafinil, Nafcillin, Nevirapine, Oxcarbazepine, Phenobarbital, Phenytoin, Primidone, Rifabutin, Rifampin, Rifapentine, St. John's wort, Sulfadimidine, Sulfinpyrazone, Troglitazone, Troleandomycin. All concomitant medications must be recorded.
* Sexually Active Patients: For all sexually active patients, the use of adequate contraception (hormonal or barrier method of birth control) will be required prior to study entry and for the duration of study participation. The non-pregnant status will be determined in all women of childbearing potential.
* Patients must have signed an approved informed consent.

Exclusion Criteria:

* Active central nervous system (CNS) disease

  a. Subjects with a history of CNS metastases or cord compression are allowable if they have been clinically stable for at least 6 weeks since completion of definitive treatment, are off steroids (if the steroids were part of the CNS disease treatment), and in the case of brain metastases, have stable or improved imaging at least 6 weeks after completion of their definitive treatment.
* Any serious medical or psychiatric illness that would prevent either the giving of informed consent or the receipt of treatment.
* Patients pregnant or nursing.
* Patients who have used tobacco or nicotine products or medications within the last three months given their significant effect on erlotinib drug levels.
* Diabetes. Defined as HgbA1C ≥ 6.5%.
* Prior metformin treatment OR EGFR targeted therapy.
* Rapidly progressive disease as judged by the investigator (Examples include rapidly deteriorating performance status or symptomatic lymphangitic spread).
* Patient has any condition associated with increased risk of metformin-associated lactic acidosis (e.g. congestive heart failure defined as New York Heart Association (NYHA) Class III or IV functional status, history of acidosis of any type; habitual intake of 3 or more alcoholic beverages per day).

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose of metformin in combination with a fixed dose of 150 mg erlotinib daily | Up to 5 weeks
  The highest dose of a treatment that does not cause unacceptable side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kalinsky, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided